CLINICAL TRIAL: NCT06882616
Title: The Effect of Laparoscopic Sleeve Gastrectomy on the Change in Carotid Intima-media Thickness in Patients With Obesity: Prospective Randomized Trial
Brief Title: the Change in Carotid Intima-media Thickness After Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammed Taha Demirpolat, Clinical Professor, Umraniye Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Carotis intima-media thickness
Record Dates: First submitted 2025-03-05; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Weight Loss; Reduce the Risk of Cardiac Disease; Carotis Intima-media Thickness
Keywords: Carotis intima-media thickness; Laparoscopic sleeve gastrectomy
MeSH Terms: conditions — Weight Loss | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Prospective, observational
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laparoscopic sleeve gastrectomy (Other): laparoscopic sleeve gastrectomy
  Interventions: Other: surgery

INTERVENTIONS:
Other: surgery — All patients will be perform laparoscopic sleeve gastrectomy. Carotid intima-media thickness will be analyzed preoperatively and at the end of the first postoperative year.

SUMMARY:
The aim of this study was to compare carotid intima-media thicknesses in laparoscopic sleeve gastrectomy patients preoperatively and at the end of the first postoperative year.

DETAILED DESCRIPTION:
Obesity is not only a disease in itself, but also predisposes to many other diseases. Cardiac diseases are one of the systems that obesity predisposes to. Obesity has been found to increase the risk of cardiac disease by increasing carotid intima-media thickness in patients with obesity. Surgery is known to be the most effective treatment for obesity and laparoscopic sleeve gastrectomy is the most common bariatric surgery procedure. Laparoscopic sleeve gastrectomy may reduce the risk of cardiac disease by reducing carotid intima-media thickness in patients with obesity through effective weight loss.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old,
* BMI > 35 kg/m2
* Laparoscopic sleeve gastrectomy will be performed
* patients with cardiac disease

Exclusion Criteria:

* patients without cardiac disease
* patients who performed other bariatric surgery procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
carotid intima-media thickness | From enrollment to the end of the first year after laparoscopic sleeve gastrectomy
  The primary outcome of the study was to compare carotid intima-media thickness at the end of the first postoperative year after laparoscopic sleeve gastrectomy (LSG) with baseline carotid intima-media thickness in patients with obesity. The investigators will measure carotid intima-media thickness with carotid doppler ultrasound before LSG and at the end of the first year after LSG and compare the results.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Taha Demirpolat, Assoc. Prof., Study Director — University of Health Sciences Umraniye Training and Research Hospital
Locations (1):
- Muhammed Taha Demirpolat, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators can share the results of statistical analysis